CLINICAL TRIAL: NCT04928313
Title: A Phase IV, Post-marketing, Prospective, Multicenter Study to Investigate the Safety and Effectiveness of Cinnomer® (Glatiramer-Acetate) in Multiple Sclerosis (MS) Treatment in Iran
Brief Title: Safety and Effectiveness of Cinnomer® (Glatiramer Acetate) in Multiple Sclerosis (MS) Treatment in Iran
Status: Completed | Type: Observational
Sponsor: Cinnagen (Industry)
Responsible Party: Sponsor
Other Study IDs: CINNOMER.CIN.AN.94 (IV)
Record Dates: First submitted 2021-04-14; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Glatiramer Acetate; Multiple Sclerosis; Quality of Life; Cinnomer; Annualized Relapse Rate; Safety; Relapsing
MeSH Terms: conditions — Multiple Sclerosis; Recurrence | interventions — Glatiramer Acetate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Glatiramer Acetate — Cinnomer® was injected subcutaneously 3 times per week at least 48 hours apart.
  Other Names: Cinnomer®

SUMMARY:
This trial was an obsevational phase IV prospective multicenter study designed to evaluate the safety and effectiveness of Cinnomer® in patients with MS in Iran.

The primary objective of this study was safety assessment of Cinnomer®

Secondary objectives were:

* Effectiveness assessment of Cinnomer®
* Assessment of the patients' QoL
* Evaluation of the patients' depression status

DETAILED DESCRIPTION:
This trial was an observational phase IV prospective multicenter study designed to evaluate the safety and effectiveness of Cinnomer® in patients with MS in Iran.

The primary objective of this study was safety evaluation. To evaluate the safety of Cinnomer®, at each visit, the AEs, seriousness of observed AEs, and abnormal laboratory findings were recorded.

To evaluate the effectiveness of Cinnomer® as the secondary objective, the indicative parameters of MS activity, including relapse information, MRI findings, and EDSS scores were considered. Also, questionnaires assessing the patients' QoL and depression were evaluated.

The sample size of 368 patients and the 14 months of the study was considered applicable for safety and effectiveness evaluation of Cinnomer®, 40 mg/ml, three times per week, in patients with relapsing forms of MS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with RRMS
* Patients diagnosed as SPMS with relapse
* All the patients taking other DMTs and their medication had been changed to Cinnomer® due to any reason.
* 0 ≤ EDSS ≤ 5
* 18 ≤ Age ≤ 60

Exclusion Criteria:

* History of hypersensitivity to Glatiramer Acetate, mannitol, or any component of the formulation.
* In the investigator's opinion, any reason that makes the subject unsuitable for treatment with Cinnomer®.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with relapsing forms of MS
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2015-04-12 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Safety assessment | Throughout the study period (up to 14 months for each patient)
  To evaluate the safety of Cinnomer®, in each visit, the AEs with any severities were recorded using system organ classes and preferred terms of the medical dictionary for regulatory activities (MedDRA Desktop Browser 4.0 Beta).

SECONDARY OUTCOMES:
Change from Baseline in Annualized Relapse Rate | Baseline, Month 14
  A clinical relapse is defined as new or recurrent neurological symptoms, not associated with fever, lasting for at least 24 hours, and followed by a period of 30 days of stability or improvement.
The proportion of relapse-free patients | Baseline, Month 14
  A clinical relapse is defined as new or recurrent neurological symptoms, not associated with fever, lasting for at least 24 hours, and followed by a period of 30 days of stability or improvement.
Change from Baseline in Expanded Disability Status Scale (EDSS) | Baseline, Month 14
  The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in seven functional systems on examination by a neurologist.
Change in Mean Number of T2 and Gd-enhancing lesions | Baseline, Month 14
Change From Baseline in Multiple Sclerosis International Quality of Life (MusiQoL) Questionnaire Scale Score at Month 14 | Baseline, Month 14
  A score of 0 = the worst QoL and a score of 100 = the best QoL
Change From Baseline in the Beck Depression Inventory II (BDI-II) Total Score at month 14 | Baseline, Month 14
  Depressive symptoms were measured by the BDI-II, a 21-item, self-reported rating inventory that measures characteristic attitudes and symptoms of depression

CONTACTS AND LOCATIONS:
Overall Officials: Abdorreza Naser Moghadasi, Assistant Professor, Principal Investigator — Multiple Sclerosis Research Center, Neuroscience Institute, Tehran University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided